CLINICAL TRIAL: NCT06922188
Title: Development of Measures to Screen for Financial Hardship in Alzheimer's Disease and Dementia
Acronym: AD/ADRD
Status: Recruiting | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Salene Jones, PhD, MA, Associate Professor, Fred Hutchinson Cancer Center
Other Study IDs: 20510; 1R01AG088347 (NIH); RG1124668 (Other: Fred Hutchinson Cancer Center)
Record Dates: First submitted 2025-03-18; First posted 2025-04-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Financial Hardship; Alzheimer's Disease (AD); Alzheimer's Disease and Related Dementia (ADRD)
Keywords: Social Determinants of Health; Financial Toxicity; Financial Burden; Dementia; Alzheimers Disease
MeSH Terms: conditions — Financial Stress; Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer's Disease and Related Dementias (ADRD) Financial Burden Cohort: The cohort consists of patients diagnosed with Alzheimer's Disease (AD) and related dementias (ADRD). Participants are identified based on clinical diagnostic criteria, including cognitive assessments.
  This study examines the financial burden associated with AD/ADRD from the patient's perspective.
- Caregivers of Patients with Alzheimer's Disease and Related Dementias (ADRD) Financial Burden Cohort: This cohort consists of caregivers providing care for patients diagnosed with Alzheimer's Disease (AD) and related dementias (ADRD). Caregivers may be family members, or friends who assist with financial management and other tasks such as daily activities, medical management, and decision-making.
  This study evaluates the financial burden experienced by caregivers of individuals with AD/ADRD.

SUMMARY:
Alzheimer's Disease and related dementias (AD/ADRD) are common and debilitating conditions. Financial hardship, a multidimensional construct of financial strain, financial stress and asset depletion, is common in AD/ADRD due to exorbitant out-of-pocket spending such as for long-term care, lower work productivity and income for their caregivers that can last for decades after disease onset, and difficulty deciding between nursing home care or home-based care while negotiating insurance coverage. People from historically marginalized groups can experience a double disparity with fewer financial resources to manage AD/ADRD and a greater risk of AD/ADRD. Screening for financial hardship in AD/ADRD is key for addressing the needs of patients and caregivers but critical barriers include a lack of suitable screening measures. Current measures are very general and meant for people without chronic medical conditions or are specific to other diseases. To fill this gap, this study will create a suite of measures that can screen for financial hardship in people with AD/ADRD and their families and caregivers. The measures will include a set to assess caregiver burden; a set to assess patient hardship as reported by the caregiver for patients who cannot report for themselves; and a set of patient-reported measures for patients that are able to report for themselves. To create these financial hardship screening measures, the project will conduct the following aims. Aim 1- Develop financial hardship screening measures for Alzheimer's Disease and related dementias: Using interviews with both caregivers and people with AD/ADRD, key indicators of financial hardship that are unique to AD/ADRD and the point in the lifespan in which it occurs will be identified. The ways that social and caregiver network size affect financial hardship will also be explored. Using the interviews and previous measures, preliminary measures will be created and will be reviewed by experts and a patient and caregiver advisory board. Aim 2- Create item response theory-based screening measures for financial hardship measures in Alzheimer's Disease and related dementias: Large samples of people with AD/ADRD (n=1000) and caregivers (n=1000) will be surveyed and item response theory will be used to evaluate and revise the measures and create scoring algorithms. A sample of additional caregivers matched to primary caregivers (n=400) will also be recruited to evaluate interrater reliability of the measures. Aim 3- Evaluate the financial hardship measures across patient and caregiver populations: Using the sample from Aim 2 and item response theory, we will evaluate the financial hardship screening measures across the following groups to ensure they are unbiased and reflect true differences: race/ethnicity; patient comorbidities; stage of AD/ADRD; caregiver relationship; social network size; number of caregivers; financial support provided; and caregiver's own health status (disability, comorbidities). The resulting measures will improve identification of financial hardship in AD/ADRD.

DETAILED DESCRIPTION:
This study investigates the financial hardship experienced by individuals with Alzheimer's Disease and Alzheimer's Disease-Related Dementias (AD/ADRD) and their caregivers. The research comprises qualitative interviews, content validation surveys, and quantitative data collection to assess financial stressors, caregiving costs, and coping mechanisms.

The first phase involves conducting semi-structured interviews with individuals diagnosed with AD/ADRD and their caregivers. These interviews will be conducted virtually, by phone, or in person, with most expected to take place remotely. Informed consent will be obtained either verbally or through signed documentation, as appropriate. Participants will be interviewed separately to ensure privacy, particularly in cases where both the patient and their caregiver are involved. The interview guide will explore changes in financial circumstances before and after diagnosis, general and specific aspects of financial hardship-including financial stress, financial strain, and asset depletion-contributing factors to financial hardship, strategies used to mitigate financial burdens, and the impact of financial hardship on well-being, decision-making, and care options. Additionally, the study will examine financial management practices, including the transition of financial responsibility from the patient to caregivers, as well as the role of caregivers and social networks in financial management and hardship buffering. Interviews will be recorded and transcribed, with Spanish transcripts translated into English. Participants will receive a small incentive for participation. If a caregiver or patient expresses interest in the other member of the dyad participating, they will be contacted via email or phone for potential enrollment.

Following the qualitative phase, a structured survey will be distributed to validate the relevance and applicability of financial hardship indicators identified during the interviews. Participants will receive an email with a study invitation and a survey link, where they will review definitions of financial hardship domains, assess the relevance of each survey item based on the perspective of the caregiver and patient, and provide demographic and job-related information. To optimize participant burden, randomized subsets of the survey will be assigned if the item bank is extensive. Participants will receive a small incentive for survey completion.

After eligibility screening, participants will complete a financial hardship survey either online or via mail. Online participants will review an electronic consent statement before proceeding, while mail-in participants will sign and return a consent form along with their completed survey using a prepaid return envelope. The survey will collect data on financial stressors, caregiving costs, and coping mechanisms. Participants will receive informational handouts on financial support resources and mental health care services. The study will examine financial caregiving networks and social support structures, as well as how financial hardship influences long-term care decisions and overall well-being. Participants will be compensated for their time and contribution to the study.

Quality control and data management processes will ensure the integrity and accuracy of study data. Surveys and interview transcripts will undergo validation checks to ensure data consistency. Data will be categorized using structured coding frameworks. A mixed-methods approach will be employed for analysis, using qualitative thematic analysis for interview data and statistical modeling for survey responses.

This study aims to improve the understanding of financial hardship among individuals with AD/ADRD and their caregivers, providing critical insights to inform policy interventions and support strategies for affected individuals and their families.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* One of the following:

  * Clinical diagnosis of Alzheimer's disease or related dementia
  * Being a caregiver to individuals with clinical diagnosis of Alzheimer's disease or related dementia
* Able to read and speak English or Spanish
* Able to provide informed consent
* Residing in the United States

Exclusion Criteria:

• Cognitive impairment precluding informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals with Alzheimer's Disease or Related Dementias (AD/ADRD) and financial caregivers providing financial support for AD/ADRD patients.
Sampling Method: Non-Probability Sample
Enrollment: 2460 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-09-18 (Estimated); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
Thematic Analysis of Qualitative Interviews to Inform Measure Development | Month 6 to Month 18 of the study
  Qualitative interviews with patients and caregivers will be conducted and analyzed using a framework analysis approach. Interview data will be used to refine our conceptual model of financial hardship (Jones et. al 2024). The unit of measure will be the number of major thematic categories identified through qualitative analysis and the number of conceptual domains established in the finalized model.
Internal Consistency of Financial Hardship Item Banks | At initial survey administration (approximately Month 19 to month 42 of the study)
  Internal consistency of the financial hardship item banks will be evaluated using Cronbach's alpha for each domain. The unit of measure will be the alpha coefficient (range 0-1), with higher values indicating greater internal consistency.
Construct Validity of Financial Hardship Item Banks | At initial survey administration (approximately Month 19 to month 42 of the study)
  Construct validity will be assessed by examining correlations between financial hardship scores and related constructs, such as quality of life, stress, and social connectedness. The unit of measure will be Pearson or Spearman correlation coefficients (range -1 to 1). The direction and strength of these correlations will be used to evaluate convergent validity.
Item-Level Performance Using Item Response Theory | At initial survey administration (approximately Month 19 to month 42 of the study)
  Item-level performance for each financial hardship item bank will be assessed using item response theory (IRT) modeling. The unit of measure will be the discrimination (slope) and severity (threshold) parameters, reported for each item individually.

CONTACTS AND LOCATIONS:
Overall Officials: Salene MW Jones, PhD, MA, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones SMW, Gaffney A, Unger JM. Common methods of determining meaningful change in clinical practice: implications for precision patient-reported outcomes. Qual Life Res. 2023 May;32(5):1231-1238. doi: 10.1007/s11136-022-03246-4. Epub 2022 Sep 10. PMID 36087227
- [Background] Jones SMW, Du Y, Bell-Brown A, Bolt K, Unger JM. Feasibility and Validity of Asking Patients to Define Individual Levels of Meaningful Change on Patient-Reported Outcomes. J Patient Cent Res Rev. 2020 Jul 27;7(3):239-248. doi: 10.17294/2330-0698.1742. eCollection 2020 Summer. PMID 32760755
- [Background] Jones SM, Amtmann D. Health care worry is associated with worse outcomes in multiple sclerosis. Rehabil Psychol. 2014 Aug;59(3):354-9. doi: 10.1037/a0037074. Epub 2014 Jul 14. PMID 25019308
- [Background] Jones SM, Amtmann D. Differential item function analysis of a scale measuring worry about affording healthcare in multiple sclerosis. Rehabil Psychol. 2016 Nov;61(4):430-434. doi: 10.1037/rep0000105. Epub 2016 Aug 29. PMID 27571410
- [Background] Jones SMW, Walker R, Fujii M, Nekhlyudov L, Rabin BA, Chubak J. Financial difficulty, worry about affording care, and benefit finding in long-term survivors of cancer. Psychooncology. 2018 Apr;27(4):1320-1326. doi: 10.1002/pon.4677. Epub 2018 Mar 8. PMID 29462511
- [Background] Jones SM, Henrikson NB, Panattoni L, Syrjala KL, Shankaran V. A theoretical model of financial burden after cancer diagnosis. Future Oncol. 2020 Dec;16(36):3095-3105. doi: 10.2217/fon-2020-0547. Epub 2020 Sep 25. PMID 32976048
- [Background] Jones SMW, Schuler TA, Padamsee TJ, Andersen MR. Financial Anxiety is Associated With Cancer Screening Adherence in Women at High Risk of Breast Cancer. Ann Behav Med. 2021 Nov 18;55(12):1241-1245. doi: 10.1093/abm/kaab010. PMID 33761532
- [Background] Kirchhoff A, Jones S. Financial Toxicity in Adolescent and Young Adult Cancer Survivors: Proposed Directions for Future Research. J Natl Cancer Inst. 2021 Aug 2;113(8):948-950. doi: 10.1093/jnci/djab014. No abstract available. PMID 33839777
- [Background] Jones SMW, Banegas MP, Steiner JF, De Marchis EH, Gottlieb LM, Sharp AL. Association of Financial Worry and Material Financial Risk with Short-Term Ambulatory Healthcare Utilization in a Sample of Subsidized Exchange Patients. J Gen Intern Med. 2021 Jun;36(6):1561-1567. doi: 10.1007/s11606-020-06479-6. Epub 2021 Jan 19. PMID 33469762
- [Background] Jones SM, Heffner JL. Financial anxiety: a potential new target to increase smoking cessation. Future Oncol. 2022 Mar;18(9):1035-1038. doi: 10.2217/fon-2021-1570. Epub 2022 Feb 8. No abstract available. PMID 35132901
- [Background] Jones SM, Lange J, Turner J, Cherkin D, Ritenbaugh C, Hsu C, Berthoud H, Sherman K. Development and Validation of the EXPECT Questionnaire: Assessing Patient Expectations of Outcomes of Complementary and Alternative Medicine Treatments for Chronic Pain. J Altern Complement Med. 2016 Nov;22(11):936-946. doi: 10.1089/acm.2016.0242. Epub 2016 Sep 30. PMID 27689427
- [Background] Jones SMW, Du Y, Panattoni L, Henrikson NB. Assessing Worry About Affording Healthcare in a General Population Sample. Front Psychol. 2019 Nov 22;10:2622. doi: 10.3389/fpsyg.2019.02622. eCollection 2019. PMID 31824388
- [Background] Lewis CC, Wellman R, Jones SMW, Walsh-Bailey C, Thompson E, Derus A, Paolino A, Steiner J, De Marchis EH, Gottlieb LM, Sharp AL. Comparing the performance of two social risk screening tools in a vulnerable subpopulation. J Family Med Prim Care. 2020 Sep 30;9(9):5026-5034. doi: 10.4103/jfmpc.jfmpc_650_20. eCollection 2020 Sep. PMID 33209839
- [Background] Lewis CC, Jones SMW, Wellman R, Sharp AL, Gottlieb LM, Banegas MP, De Marchis E, Steiner JF. Social risks and social needs in a health insurance exchange sample: a longitudinal evaluation of utilization. BMC Health Serv Res. 2022 Nov 28;22(1):1430. doi: 10.1186/s12913-022-08740-6. PMID 36443789
- [Background] Jones SMW, Unger JM. Tailoring Pain Interference Measurement in People with Cancer: A Feasibility Study. J Pain Symptom Manage. 2022 Jul;64(1):e35-e41. doi: 10.1016/j.jpainsymman.2022.02.334. Epub 2022 Feb 27. PMID 35235855
- [Background] Jones SMW, Ton M, Malen RC, Newcomb PA, Heffner JL. Item response theory analysis of benefits and harms of cannabis use in cancer survivors. J Natl Cancer Inst Monogr. 2024 Aug 15;2024(66):275-281. doi: 10.1093/jncimonographs/lgad022. PMID 39108240
- [Background] Noel PH, Jones S, Parchman ML. Patient Experience in an Era of Primary Care Transformation: Revisiting the PACIC. Eur J Pers Cent Healthc. 2016;4(3):528-540. PMID 27746917
- [Background] Jones SMW, Yi JC, Jim HSL, Loren AW, Majhail NS, Uberti J, Whalen V, Leisenring WM, Flowers MED, Lee SJ, Syrjala KL. Age and gender differences in financial distress among hematopoietic cell transplant survivors. Support Care Cancer. 2020 Sep;28(9):4361-4371. doi: 10.1007/s00520-019-05291-1. Epub 2020 Jan 8. PMID 31916007
- [Background] Jones SM, Yi J, Henrikson NB, Panattoni L, Shankaran V. Financial hardship after cancer: revision of a conceptual model and development of patient-reported outcome measures. Future Sci OA. 2024 May 14;10(1):FSO983. doi: 10.2144/fsoa-2023-0229. eCollection 2024. PMID 38827796
- See also: Research Portfolio Online Reporting Tools — https://reporter.nih.gov/search/_eom1eFaakaw--lQhfO75A/project-details/10953849

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT06922188/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT06922188/ICF_001.pdf